## **COVER PAGE**

Study title: The Feasibility and Effect of Digital Cognitive Training in Mild

Cognitive Impairment

NCT ID: Not yet assigned

**Document type:** Consent form

Original date of the document: October 30, 2023

## Consent form for participation in a health research project

Study title: "The Feasibility and Effect of Digital Cognitive Training in Mild Cognitive Impairment"

## **Declaration from the participant:**

Danish project identification no.: <u>N2023-0020</u>

I have received written and oral information about the study, and I know enough about the study's purpose, methods, time frame, and possible risks or side effects to be able to consent to participate herein.

I know that it is voluntary to participate and that I can always withdraw my consent without having to state a reason and without losing my current or future treatment rights.

I hereby consent to participate in the study and have received a copy of this consent form as well as a copy of the written study material.

| Name: |
|---|
| Date: Signature: |
| Do you want to be informed of the study's results as well as any consequences for you? Yes (put an x) No (put an x) |
| Declaration from the person giving the information: |
| I declare that the participant has received written and oral information about the study, has had opportunities to ask questions, and has been given sufficient time to consider if he or she wishes to participate herein. |
| The participant has been thoroughly informed of his or her rights, including the right to withdraw from the study without having to give a reason and without losing their current or future treatment rights. |
| The participant has been given a copy of the written study material and a copy of this consent form for their personal use. |
| Name: |
| Date:Signature: |